CLINICAL TRIAL: NCT00585507
Title: A Phase II Multi-Center Study to Evaluate the Efficacy and Safety of 500mg of Fulvestrant (Faslodex) as a First Line Hormonal Treatment in Postmenopausal Women With Hormone Receptor Positive Metastatic Breast Cancer
Brief Title: Efficacy and Safety of 500mg of Fulvestrant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Lowell General Hospital (Other); University of Colorado, Denver (Other); University of Maryland Greenebaum Cancer Center (Other); South Shore Hospital (Other)
Responsible Party: Principal Investigator, Steven Come, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-016
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: hormone receptor positive breast cancer; Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- single (Experimental): fulvestrant 500mg
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — 500mg into the muscle on days 1, 15 and 29 and then every 28 days thereafter.
  Other Names: Faslodex

SUMMARY:
Fulvestrant has proven effective in the treatment of hormone receptor positive metastatic breast cancer. The dose used in studies so far has been well tolerated and may be too low for optimal effectiveness. In this study, a higher dose will be used to see whether an improved outcome will result.

DETAILED DESCRIPTION:
* Fulvestrant will be administered by intramuscular injection on day 1, day 15 and day 29 and then every 28 days thereafter.
* Participants will have a physical examination and blood work performed on each treatment date. After teh study treatment has been completed, the physical examinations will be done every three months for the first 2 years, every 6 months for years 2-5, and annually after 5 years.
* Participants may remain on study treatment until disease progression or until they experience serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Histologically confirmed adenocarcinoma of the breast progressing local-regional or metastatic disease that is not considered amenable to curative treatment
* Evidence of hormone sensitivity of primary or secondary tumor tissue
* Postmenopausal as defined by criteria listed in protocol
* May have had adjuvant endocrine therapy if discontinued at least 12 months prior to inclusion. Subjects who have had minimal exposure to adjuvant or first line metastatic endocrine treatment during the 12 months prior to study enrollment can be eligible with overall PI and sponsor permission
* Prior trastuzumab and biologic therapy is allowed, but must be discontinued more than 2 weeks prior to inclusion
* Presence of measurable or evaluable, nonmeasurable, disease. Any x-rays and scans for assessment of measurable disease must be performed with 28 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2

Exclusion Criteria:

* Presence of life-threatening metastatic disease
* Endocrine therapy the advanced disease setting
* Systemic chemotherapy, whether as adjuvant therapy or for advanced disease, within previous 4 weeks
* Trastuzumab or biologic therapy within previous 2 weeks
* Extensive radiation therapy within the last 2 weeks
* Prior adjuvant or neoadjuvant treatment with fulvestrant is not allowed
* Concomitant anticancer treatments
* Chronic bisphosphonates for hypercalcemia or prevention of bone metastases
* Subjects receiving long-term anticoagulant therapy with warfarin
* Estrogen replacement therapy within 6 months of trial entry
* Previous or current systems malignancy within the past 3 years
* Treatment with non approved or investigational drug within 2 weeks before study entry
* Any evidence of severe or uncontrolled systemic disease
* History of bleeding diathesis
* Any severe concomitant condition which makes it undesirable for the subject to participate in the study or which would jeopardize compliance with the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-04 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical benefit rate for subjects receiving this dose and schedule of fulvestrant.

SECONDARY OUTCOMES:
Overall objective response rate, time to response, duration of response, duration of clinical benefit, and time to progression.
Assessment of adverse events | 4 years
Assessment of pharmacokinetics of this dose and schedule of fulvestrant. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Come, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (5):
- United States (5):
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - South Shore Hospital, South Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: No